CLINICAL TRIAL: NCT05120791
Title: Health-promoting Effects of the Microalga Phaeodactylum Tricornutum - Bioavailability and Excretion of Nutrients in Relation to Age and Their Effects on Fatty Acid Status and Inflammatory Markers".
Brief Title: Age Related Effects Consuming Phaeodactylum Tricornutum
Acronym: MIA_E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Professor, University of Hohenheim
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MIA_E
Record Dates: First submitted 2021-10-26; First posted 2021-11-15 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Aging; Well Aging
Keywords: Microalgae; omega-3 fatty acids; Micronutrients; carotinoids; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: 4 arm parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1,3g)
  Interventions: Dietary Supplement: Placebo vegetable bouillon
- Microalgae phaeodactylum (Active Comparator): 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1.3g), 2.3g Microalgae Phaeodactylum
  Interventions: Dietary Supplement: microalgae phaeodactylum
- Beta-Glucan (Active Comparator): 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1.3g), Beta-Glucan (1.8g)
  Interventions: Dietary Supplement: From the Microalgae phaeodactylum the extracted beta-Glucan (especially chrysolaminarin)
- Combi Microalgae phaeodacytlum and Beta-Glucan (Active Comparator): 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1.3g), 2.3g Microalgae, Beta-Glucan (1.8g)
  Interventions: Dietary Supplement: A combination of the vegetable bouillon, the microalgae and the beta-Glucan

INTERVENTIONS:
Dietary Supplement: Placebo vegetable bouillon — 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1,3g)
  Arms: Placebo
Dietary Supplement: microalgae phaeodactylum — 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1.3g), 2.3g Microalgae Phaeodactylum
  Arms: Microalgae phaeodactylum
Dietary Supplement: From the Microalgae phaeodactylum the extracted beta-Glucan (especially chrysolaminarin) — 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1.3g), Beta-Glucan (1.8g)
  Arms: Beta-Glucan
Dietary Supplement: A combination of the vegetable bouillon, the microalgae and the beta-Glucan — 14 days wahs-out: no fish eating 14 days: no fish eating, the participants eat vegetable bouillon (1.3g), 2.3g Microalgae, Beta-Glucan (1.8g)
  Arms: Combi Microalgae phaeodacytlum and Beta-Glucan

SUMMARY:
Investigation of the microalgae Phaeodactylum as food with regard to the uptake of omega-3 fatty acids and effects on various blood parameters in relation to age.

Bioavailability and excretion of nutrients and their effects on fatty acid status and inflammatory markers.

DETAILED DESCRIPTION:
Due to a multifaceted redesign of all areas of life, older people face many nutritional challenges, such as cognitive change, sarcopenia and micronutrient deficiency. In addition to age-associated diseases, cognitive decline is usually a precursor to neurodegenerative processes, such as Alzheimer's disease. The full molecular mechanisms are still unknown, but classic aging mechanisms, such as oxidative stress and subclinical inflammation, play a role. Due to the changed life situation, there is a reduced need for energy, while the need for nutrients remains, which greatly increases the risk of malnutrition in old age. This results in an increasing prevalence of sarcopenia. The decrease in muscle mass and strength leads to functional limitations in the elderly and also promotes oxidative stress. This increases the need for antioxidant nutrients such as carotenoids and vitamins. Studies show that age-related chronic subclinical inflammation, such as occurs in the context of an omega-6 fatty acid (-FS) emphasized diet, plays a central role in the pathogenesis of age-associated diseases

Due to this, the microalgae PT could be a goud supplier of nutrients like omega-3 FS, especially eicosapentaenoic acid (EPA), which is otherwise found mainly in fatty fish, and Fucoxanthin, an antioxidant. The investigator study the change of omega-3, -6 and -9 FS in blood plasma, in erythrocytes, as well as the change of fucoxanthin and beta-carotene. The investigator measure blood parameters for safety and control the influence on the intestinal barrier.

ELIGIBILITY:
Inclusion Criteria:

Age ≥60 ≤90 years, weight ≥50 kg, generally healthy

* Signed informed consent form
* Willingness to follow the prescribed diet for the duration of the study
* No participation in any other clinical trial (current or within the last 30 days)

Exclusion Criteria:

* Taking intestinal therapeutics, antibiotics, immunosuppressants or similar. (if necessary, decision on a case-by-case basis)
* Pregnancy/breastfeeding
* Relevant violations of the dietary protocol
* Occurrence of relevant diseases (if necessary, individual case decision)
* Withdrawal of consent
* Placement in a clinic or similar facility due to official or court order

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in omega-6/omega-3 ratio (plasma level basis) | 14 days
  fatty acid chromatographic measurement

SECONDARY OUTCOMES:
Omega-3 fatty acid index | 14 days
  fatty acid chromatographic measurement in red blood cells
Uptake of fucoxanthin and beta-carotene | 14 days
  chromatographic measurement in plasma
Inflammation (CRP) | 14 days
  measurement in blood serum

OTHER OUTCOMES:
Markers for oxidative stress | 14 days
  lipid hydroperoxides)
Albumin | 14 days
  Measurement in serum
weight | 14 days
  in kilograms
FFQ- Food frequence questionnaire | 4 weeks
  Food questionnaire about the general eating of the last 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Stephan C. Bischoff, Prof. Dr, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided